CLINICAL TRIAL: NCT01510665
Title: Magnesium Supplementation in the Second Trimester of Pregnancy for Overweight Individuals
Brief Title: Magnesium Supplementation in the Second Trimester of Pregnancy to Overweight and Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Simin Liu, Dr., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Magnesium123
Record Dates: First submitted 2011-12-23; First posted 2012-01-16 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Gestational Diabetes; Obesity
Keywords: Weight gain in pregnancy; Metabolic and Inflammatory markers
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Gestational Weight Gain | interventions — magnesium citrate; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium Supplement (Experimental): Magnesium citrate dietary supplement (300 mg elemental Magnesium daily dose) given week 13 to week 28 (two pills daily)
  Interventions: Dietary Supplement: Magnesium citrate
- Placebo (Placebo Comparator): Identical appearing pill with inactive ingredients given week 13 to week 28 (two pills daily)
  Interventions: Dietary Supplement: Placebo
- Diet (Active Comparator): Nutritionist counseling session and advice on following a magnesium rich diet from week 13 to week 28
  Interventions: Behavioral: Dietary modification

INTERVENTIONS:
Dietary Supplement: Magnesium citrate — Magnesium citrate tablets 950 mg, two pills once daily (Total daily dose of 300 mg elemental magnesium)
  Arms: Magnesium Supplement
Dietary Supplement: Placebo — Identical appearing placebo with inactive ingredients, two pills once daily.
  Arms: Placebo
Behavioral: Dietary modification — Nutritionist counseling session and advice on following a magnesium rich diet
  Arms: Diet

SUMMARY:
This is a prospective, randomized, placebo controlled study with three parallel arms examining the effects of magnesium supplementation in the second trimester of pregnancy.

Recent research has shown that supplemental magnesium can have beneficial effects, especially in overweight individuals. Not only do many people have a magnesium deficient diet, there is also evidence that magnesium can improve blood sugar levels. Due to the growing concern of obesity with pregnancy and its associated complications, such as diabetes and abnormal fetal growth, magnesium therapy could have novel and beneficial effects on pregnancy outcomes.

In this study, 60 overweight and obese pregnant patients in their first trimester will be enrolled and randomized. The first group (A) will receive oral magnesium citrate (300mg elemental Magnesium), group B will receive dietary counseling about following a magnesium rich diet from a nutritionist, and group C will receive a placebo (control). Blood and urine specimens will be collected at three time points during the pregnancy to analyze changes in levels of metabolic markers, inflammatory markers, and protein expression profiles. Fetal and maternal complications of pregnancy will be noted, including maternal weight gain. At delivery, patients will have a placental cord blood specimen and placental biopsy collected for gene expression patterns and further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age
* Pregnant in the first trimester
* Able to give informed consent
* Planning to deliver at UCLA
* BMI greater than or equal to 25

Exclusion Criteria:

* On insulin therapy or other oral hypoglycemic agents
* Multiple gestation
* Baseline HgbA1C > 6.5%
* Prior history of clinically diagnosed T2D
* Multiple dietary restrictions/food allergies
* Heart, renal, or liver failure
* Clinical history of psychiatric illness or substance abuse
* Out of town travel planned at study visits

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in maternal biomarkers during pregnancy up to 28 weeks | up to 28 weeks
  Blood and urine markers of inflammatory and metabolic markers will be assessed during the pregnancy,comparing baseline values to second trimester values, which will be up to 28 weeks.
Neonatal birth weight/height | Up to 10 months
  This measure will be assessed at neonatal delivery, which will occur at a maximum of up to 10 months from randomization. Neonatal weight and height at birth will be assessed.
Change in maternal biomarkers in pregnancy in the third trimester | Up to 36 weeks
  Blood and urine markers of inflammatory and metabolic markers will be assessed during the pregnancy,comparing baseline values to third trimester values, which will be up to 36 weeks.

SECONDARY OUTCOMES:
Neonatal outcomes | Up to 10 months
  This measure will be assessed at neonatal delivery, which will occur at a maximum of up to 10 months from randomization. At delivery, neonatal characteristics will be assessed:
  Macrosomia, preterm birth, head circumference, and apgar score.
Neonatal tertiary outcomes | Up to 10 months
  This measure will be assessed at neonatal delivery, which will occur at a maximum of up to 10 months from randomization. Cord blood and placenta will be collected at delivery, and we will examine endothelial progenitor cell presence in cord blood, PON expression in cord blood, and DNA expression from the placental tissue.
Pregnancy complications | Up to 10 months
  From date of randomization until the date of delivery of the neonate, up to a maximum of 10 months, pregnancy complications such as development of gestational diabetes, hypertension, proteinuria, shoulder dystocia, cesarean section, as well as amount of weight gain will be assessed from the chart.

CONTACTS AND LOCATIONS:
Overall Officials: Simin Liu, MD, ScD, MS, MPH, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - 200 Medical Plaza UCLA Ob/Gyn Clinic, Westwood, Los Angeles, California
  - West Medical UCLA Ob/Gyn Clinic, Westwood, Los Angeles, California